CLINICAL TRIAL: NCT05028465
Title: The Efficacy and Safety of Endoscopic Papillectomy Combined With Endobiliary Radiofrequency Ablation for Ampullary Neoplasms With Intraductal Biliary Extension
Brief Title: EP Combined With RFA for Ampullary Neoplasms With Intraductal Biliary Extension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Professor, First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-08-118
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Ampullary Adenomas
Keywords: Endoscopic papillectomy; Radiofrequency ablation; Ampullary neoplasms; Intraductal biliary extension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EP combined with RFA (Experimental): Endoscopic Papillectomy Combined with Endobiliary Radiofrequency Ablation
  Interventions: Procedure: Endoscopic Papillectomy; Procedure: Endobiliary Radiofrequency Ablation

INTERVENTIONS:
Procedure: Endoscopic Papillectomy — A snare devicewas inserted via the working channel, and the endoscopist adjusted the snare to securely grasp the lesion, which was then excised by using standard electrocautery.
Procedure: Endobiliary Radiofrequency Ablation — The RFA catheter was then placed under fluoroscopic guidance across the distal common bile duct. An ERBE VIO200D generator (ERBE Elktromedizin, Tubingen, Germany) was connected for RFA at 10 W for 90 seconds.

SUMMARY:
Endoscopic papillectomy is the preferred approach for management of ampullary adenomas. Endobiliary radiofrequency ablation (RFA) is an ablative therapy that has been used to treat malignant biliary strictures. The aim of this study was to evaluate the safety and efficacy of endoscopic papillectomy combined with endobiliary RFA for ampullary neoplasms with intraductal biliary extension.

DETAILED DESCRIPTION:
Ampullary neoplasms remain rare, with a reported prevalence of 0.04% to 0.12% in autopsy studies. , endoscopic papillectomy is now recognized as a safe and reliable alternative to surgery for ampullary adenomas and is associated with high success rates (72%-95%), low morbidity (10%-30%), and minimal mortality (0.2%-1%). Typically, however, intrabiliary extension of the adenoma has been regarded as a contraindication for endoscopic papillectomy. Surgical referral is therefore recommended with intraductal extension, particularly when the length of extension exceeds 1 cm. Radiofrequency ablation offers a potentially safe and effective treatment for malignant biliary strictures. The use of RFA as a primary treatment for intraductal dysplasia after endoscopic papillectomy has been shown in few small case series to be feasible with the primary limitation of short follow-up periods. The primary aim of this study was to describe our experience with RFA in patients with ampullary neoplasia and associated intraductal extension who were not surgical candidates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven ampullary adenoma or adenocarcinoma with intraductal biliary extension ≥1cm who were deemed medically unfit for surgery or declined surgery

Exclusion Criteria:

* pancreatic invasion, lymph node invasion, distant metastasis, or coagulopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02-10 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Recurrence | one year
  Recurrence was defined as discovery of neoplasia after a negative surveillance endoscopy and biopsy

SECONDARY OUTCOMES:
Complete resection of ampullary adenomas | three months
  Complete resection of ampullary adenomas was confirmed when no residual tissue was found on ampullary and intraductal biopsies at the 3-month follow-up ERCP.
Endoscopic success | six months
  Endoscopic success was defined as complete ablation of the lesion without residual neoplasia or recurrence at the 6-month follow-up endoscopy.
adverse events | one months
  adverse events such as bleeding, acute pancreatitis after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, Dr., Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson RR, Muthusamy VR. Radiofrequency ablation for intraductal extension of ampullary neoplasms: Are we ready to feel the burn? Gastrointest Endosc. 2017 Jul;86(1):177-179. doi: 10.1016/j.gie.2016.12.022. No abstract available. PMID 28610856
- [Background] Camus M, Napoleon B, Vienne A, Le Rhun M, Leblanc S, Barret M, Chaussade S, Robin F, Kaddour N, Prat F. Efficacy and safety of endobiliary radiofrequency ablation for the eradication of residual neoplasia after endoscopic papillectomy: a multicenter prospective study. Gastrointest Endosc. 2018 Sep;88(3):511-518. doi: 10.1016/j.gie.2018.04.2332. Epub 2018 Apr 13. PMID 29660322
- [Background] Yang J, Wang J, Zhou H, Zhou Y, Wang Y, Jin H, Lou Q, Zhang X. Efficacy and safety of endoscopic radiofrequency ablation for unresectable extrahepatic cholangiocarcinoma: a randomized trial. Endoscopy. 2018 Aug;50(8):751-760. doi: 10.1055/s-0043-124870. Epub 2018 Jan 17. PMID 29342492